CLINICAL TRIAL: NCT04300036
Title: Efficacy and Safety of Longan Syrup in Healthy Volunteers With Insomnia
Acronym: longan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 829/62
Record Dates: First submitted 2020-02-24; First posted 2020-03-09 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Insomnia
Keywords: longan; insomnia; efficacy; safety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- longan syrup (Experimental): Take 15 ml of longan syrup once a day for 3 months
  Interventions: Dietary Supplement: longan syrup
- Placebo syrup (Placebo Comparator): Take 15 ml of placebo syrup once a day for 3 months
  Interventions: Dietary Supplement: Placebo syrup

INTERVENTIONS:
Dietary Supplement: longan syrup — Subjects will take 15 ml of longan syrup once a day for 3 months
  Arms: longan syrup
Dietary Supplement: Placebo syrup — Subjects will take 15 ml of placebo syrup once a day for 3 months
  Arms: Placebo syrup

SUMMARY:
The objectives of this study were to evaluate efficacy and safety of longan syrup in healthy volunteers with insomnia. Subjects will take 15 ml of longan syrup once a day for 3 months. They will be investigated their insomnia using Insomnia Severity Index (ISI) questionnaire, Thai- The Pittsburgh Sleep Quality Index (PSQI) questionnaire,STOP - BANG questionnaire, Epworth Sleepiness Scale (ESS) questionnaire, Actiwatch, plasma cortisol, aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), creatinine (Cr), blood urea nitrogen (BUN), fasting blood sugar, HbA1C, complete blood count (CBC), hemoglobin, lipid profile, phosphate level, saliva cortisol, and urine melatonin before and after taken longan syrup.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-65 years
* Insomnia severity index (ISI) more than 7
* Thai- The Pittsburgh Sleep Quality Index (PSQI)) more than 5
* STOP - BANG less than 5
* No diabetes mellitus and thyroid dysfunction
* Fasting plasma glucose less than 126mg/dl
* Can communication (reading and writing)
* Be willing to be subjects in this study

Exclusion Criteria:

* Know longan allergy or have history of adverse events from longan
* Take benzodiazepine, melatonin, valerian, and St Johns Wort in 1 month before this study starting
* Take medicines, herbs, or food supplements including thiazide diuretics, beta-blockers ,and estrogen that have an effect on blood sugar level in 1 month before this study starting
* Cannot control comorbidity diseases
* Irregular working hours
* Pregnancy or breast feeding
* Participated in other studies

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-02-10 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index | 3 months
  Insomnia severity index after taken longan syrup will be less than before taken. The minimum and maximum values are 0 and 28 scores, respectively. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Thai- The Pittsburgh Sleep Quality Index | 3 months
  Thai- The Pittsburgh Sleep Quality Index after taken longan syrup will be less than before taken. The minimum and maximum values are 0 and 21 scores, respectively. Higher scores mean a worse outcome.
Snoring, Tiredness, Observed apnea, blood Pressure, Body mass index, Age, Neck circumference and Gender questionaire | 3 months
  Snoring, Tiredness, Observed apnea, blood Pressure, Body mass index, Age, Neck circumference and Gender questionaire (STOP - BANG) after taken longan syrup will not be more than before taken. The minimum and maximum values are 0 and 8 scores, respectively. Higher scores mean a worse outcome.
Epworth sleepiness scale | 3 months
  Epworth sleepiness scale after taken longan syrup will be less than before taken. The minimum and maximum values are 0 and 24 scores, respectively. Higher scores mean a worse outcome.
Actiwatch value | 3 months
  Actiwatch value after taken longan syrup will be better than before taken.
Serum cortisol | 3 months
  Serum cortisol value at 8.00 o'clock (normal value 5-23 mcg/dL) after taken longan syrup will not be less than before taken.
Saliva cortisol | 3 months
  Saliva cortisol at 20.00 o'clock (normal value 3.9 +/- 0.2 nmol/L (range 2.2-4.1 nmol/L)) after taken longan syrup will not be more than before taken.
Urine Melatonin | 3 months
  Urine Melatonin overnight (in ng/mL) after taken longan syrup will not be less than before taken.
Serum Low-density lipoprotein | 3 months
  Serum Low-density lipoprotein (in mg/dL) after taken longan syrup will not be more than before taken.
Serum High-density lipoprotein | 3 months
  Serum High-density lipoprotein (in mg/dL) after taken longan syrup will not be more than before taken.
Serum total cholesterol | 3 months
  Serum total cholesterol (in mg/dL) after taken longan syrup will not be more than before taken.
Serum triglyceride | 3 months
  Serum triglyceride (in mg/dL) after taken longan syrup will not be more than before taken.
Glycohemoglobin | 3 months
  Glycohemoglobin (Hemoglobin A1c) (in %) after taken longan syrup will not be more than before taken.
Fasting plasma glucose | 3 months
  Fasting plasma glucose (in mg/dL) after taken longan syrup will not be more than before taken.
Aspartate aminotransferase in serum | 3 months
  Aspartate aminotransferase (in U/L ) after taken longan syrup will not be more than before taken.
Alanine aminotransferase in serum | 3 months
  Alanine aminotransferase (in U/L ) after taken longan syrup will not be more than before taken.
Alkaline phosphatase in serum | 3 months
  Alkaline phosphatase (in U/L ) after taken longan syrup will not be more than before taken.
Serum creatinine | 3 months
  Serum creatinine (in mg/dl ) after taken longan syrup will not be more than before taken.
Blood Urea Nitrogen | 3 months
  Blood Urea Nitrogen (in mg/dl ) after taken longan syrup will not be more than before taken.
Hemoglobin | 3 months
  Hemoglobin (in g/dl ) after taken longan syrup will not be more than before taken.
Phosphate level | 3 months
  Phosphate level (in g/dl ) after taken longan syrup will not be more than before taken.
Complete blood count | 3 months
  Complete blood count (in 10^6 cells/mcl ) after taken longan syrup will not be more than before taken.

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Ph.D, Principal Investigator — Chulalongkorn University
Locations (1):
- Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn Unviersity, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No